CLINICAL TRIAL: NCT01828606
Title: Randomised Controlled Trial to Compare the Influence of Sub-bandage Pressure on Percentage Volume Reduction of Leg Lymphoedema
Brief Title: Comparative Trial to Monitor Interface Pressure in Relation to Volume Change in Leg Lymphoedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nij Smellinghe Hosptial (Other)
Responsible Party: Principal Investigator, R.J. Damstra, MD PhD, Nij Smellinghe Hosptial
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NS6NL; CLIN-PROT-EU-05-184776 (Other Grant/Funding Number: 3M Deutschland GmbH)
Record Dates: First submitted 2013-04-07; First posted 2013-04-10 (Estimated); Last update posted 2015-02-10 (Estimated); Status verified 2014-02

CONDITIONS: Lymphedema
Keywords: leg lymphedema; volume measurement; compression therapy; interface pressure; static stiffness index (SSI); volume change
MeSH Terms: conditions — Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coban 2 system (Experimental): The two layer system is more stiff and the material is different designed
  Interventions: Device: coban 2 system; Device: coban lite system
- coban lite systems (Experimental): All centres will perform the pressure measurements with Picopress, Microlab Elettronica, Italy For mobility measurements all centres will be supplied with pedometers. For perometry the centres will use their own equipment
  According to protocol the materials are applied to the whole leg and the measuring devices are put in place
  Interventions: Device: coban 2 system; Device: coban lite system

INTERVENTIONS:
Device: coban 2 system — All centres will perform the pressure measurements with Picopress, Microlab Elettronica, Italy For mobility measurements all centres will be supplied with pedometers. For perometry the centres will use their own equipment
  According to protocol the materials are applied to the whole leg and the measuring devices are put in place
Device: coban lite system — All centres will perform the pressure measurements with Picopress, Microlab Elettronica, Italy For mobility measurements all centres will be supplied with pedometers. For perometry the centres will use their own equipment
  According to protocol the materials are applied to the whole leg and the measuring devices are put in place

SUMMARY:
Although there is no doubt about the need for compression therapy in lymphoedema, it is not investigated in much detail how much pressure is needed to get optimum volume reduction. New research suggests that there is obviously an upper pressure limit beyond further increase of pressure seems contra productive. This upper limit is around 30-40 mm Hg of initial pressure exerted by inelastic bandages on the upper and around 50-60 mm Hg on the lower extremity. This study is designed to investigate the effect of pressure on %volume reduction of leg lymphoedema with 2 bandages which are very comparable in product properties (slippage, stiffness, etc.), but differ in their pressure exerted to the limb.

DETAILED DESCRIPTION:
Lymphoedema is a chronic swelling caused by the regional accumulation of protein-rich fluid in tissues due to a compromised lymphatic system. This may present as primary lymphoedema, defined as congenital abnormality of lymphatic vessels or secondary lymphoedema, acquired from various insults to the lymphatic system, such as malignancy, trauma, surgery or irradiation. It is most frequently seen after lymph node dissection, surgery or radiation therapy during cancer treatment, most notably breast cancer. In the United Kingdom a large prevalence study was undertaken by Moffatt et al and a rate of 1.33 per 1000 population was identified. In general, the prevalence increases with age and is higher in women than in men. One function of the lymphatic system is to remove fluid from the interstitial tissues and return it to the venous circulation. compression therapy is the cornerstone in the treatment of lymphoedema

Much of evidence how compression works is based on research in venous disease, which has been extrapolated to lymphoedema. Hence, compression bandaging systems available in the market are used for the treatment of venous disease and at the same time lymphoedema.

This upper limit is around 30-40 mm Hg of initial pressure exerted by inelastic bandages on the upper and around 50-60 mm Hg on the lower extremity. This is also stated in the International Lymphoedema Framework position document "Compression Therapy: A position document on compression bandaging".

100 subjects with leg lymphoedema will be enrolled into the study. The duration of study will be one week for each participant. All participants will receive compression therapy with 3M Coban 2 and 3M Coban 2 Lite respectively according to the randomisation list. The goal of the present study is to gain information on %volume reduction of lymphoedematous legs in relation to pressure.

ELIGIBILITY:
Inclusion Criteria:

1. Mobile males or females, age 18 years or older
2. Subject is mobile and able to walk minimum 5000 steps
3. Subject has unilateral or bilateral leg lymphoedema of primary or secondary origin
4. Maximum leg circumference at C position is 60 cm or less
5. Subject has more or equal than 5 mm pitting leg lymphoedema diagnosed as stage II or late stage II according to the International Society of Lymphology staging
6. Subject requires intense bandaging therapy
7. ABPI >= 0.8
8. Willing to give written informed consent and willing to comply with the study protocol

Exclusion Criteria:

1. Known pregnancy
2. Evidence of active cancer with potential or known risk of metastasis
3. Cancer treatments (surgery, chemotherapy, radiotherapy) not completed at least 6 months prior to randomisation
4. Lobes, that a proper bandage application is not possible
5. Lobes in the area where a pressure sensor needs to be placed
6. A period of intense daily bandaging within the last month
7. Any oedema not directly related to lymph failure (e.g. related to heart, renal disease etc.)
8. Diuretic treatments
9. Paralysis or neuropathy of the legs
10. Clinical infection of the legs (e.g. erysipelas)
11. Postthrombotic syndrome and/or medical conditions that are contraindicated for compression therapy
12. History of allergic reactions to study material
13. Participation in any other prospective clinical study that can potentially interfere with this study
14. Participants who are, in the opinion of the clinical investigator, unsuitable for enrolment in this study, for reasons not specified in the exclusion criteria.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-04; Primary Completion 2014-03 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
volume decrease in relation to pressure application of two types of bandages | 1 week, 2 bandages changes
  At each of the 8 visits the supine and standing pressure under the bandage is measured with a Picopress device at the B1, C and F positions. The patient will receive new bandaging twice a week. At those visits the volume is determined and a second pressure measurement is conducted 2 hours after bandage application. For safety assessment all adverse events will be documented.
  The total number of bandage changes could increase if bandage changes are required more often. On these occasions all measurements, which are required on a regular bandage change day, will be performed.

SECONDARY OUTCOMES:
pressure drop profiles under 2 bandage types | 1 week
  At each of the 8 visits the supine and standing pressure under the bandage is measured with a Picopress device at the B1, C and F positions. The patient will receive new bandaging twice a week. At those visits the volume is determined and a second pressure measurement is conducted 2 hours after bandage application. For safety assessment all adverse events will be documented.
  The total number of bandage changes could increase if bandage changes are required more often. On these occasions all measurements, which are required on a regular bandage change day, will be performed.

CONTACTS AND LOCATIONS:
Overall Officials: RJ Damstra, MD PhD, Principal Investigator — Nij smellinghe hospital, Netherlands; FJ Schingale, MD PhD, Principal Investigator — Lympho-Opt GmbH, Germany; H Partsch, MD PhD, Study Chair — professor with eremite, Austria; T Karlsmark, MD PhD, Principal Investigator — Bispebjerg Hospital, Denmark
Locations (3):
- Dermato-venerologisk afd. og videncenter for sårheling D/S Bispebjerg Hospital, København NV, Denmark
- Lympho-Opt GmbH, Pommelsbrunn, Germany
- Nij Smellinghe hospital, Drachten, Provincie Friesland, Netherlands

REFERENCES:
- See also: The foundation related to the expert centre organizing research — http://www.slcn.nl
- See also: General website form the Nij Smellinghe hospital — http://www.nijsmellinghe.nl